CLINICAL TRIAL: NCT01219998
Title: Evaluation of the Predictive Ability of Urinary NGAL as an Early Marker of Acute Kidney Injury Following Cardiac Surgery in Neonates and Infants
Brief Title: NGAL, an Early Predictive Marker of Acute Kidney Injury After Cardiac Surgery in Neonates and Infants
Acronym: NGAL
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: CRC08103; K080602 (Other: AP-HP)
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Peritoneal Lesion
Keywords: Postoperative Complications; Acute Kidney Failure; Peritoneal Dialysis; NGAL
MeSH Terms: conditions — Postoperative Complications; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples are collected during the early postoperative period, stored, than NGAL concentrations are measures on the ARCHITECT platform.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NGAL Kinetics in neonates: to describe postoperative kinetics of urinary NGAL in neonates and to identify the threshold for accurate prediction of severe AKI requiring RRT in neonates and infants undergoing cardiac surgery with cardiopulmonary bypass

SUMMARY:
Urinary NGAL has been shown to be an early marker of acute kidney injury (AKI) following paediatric cardiac surgery (2 hours off pump). Previous studies showed that an early increase of urinary NGAL following cardiopulmonary bypass was predictive of AKI. Several studies included heterogeneous populations of children undergoing cardiac surgery, but NGAL has not been studied in neonates after open heart surgery, neither has been identified the threshold for accurate prediction of severe AKI requiring renal replacement therapy.

The aim of this observational cohort study is to describe postoperative kinetics of urinary NGAL in neonates and to identify the threshold for accurate prediction of severe AKI requiring renal replacement therapy in neonates and infants undergoing cardiac surgery

DETAILED DESCRIPTION:
Urinary NGAL has been shown to be an early marker of AKI following paediatric cardiac surgery (2 hours off pump). Previous studies showed that an early increase of urinary NGAL following cardiopulmonary bypass was an excellent predictor for a later >50% increase in serum creatinine concentration in children undergoing cardiac surgery. Increased urinary concentrations of NGAL were found following open heart surgery. When defining AKI as an >50% increase of serum creatinine from baseline, the increase of urinary NGAL concentration two hours off pump appeared to be an excellent predictor of AKI. Several studies included heterogeneous populations of patients aged one month to 21 years undergoing cardiac surgery. Besides, NGAL concentrations have not been studied in neonates after open heart surgery, neither has been identified the threshold for accurate prediction of severe AKI requiring renal replacement therapy (RRT). If such a threshold was identified, urinary NGAL could be provided for intervention.

The aim of this observational cohort study is to describe postoperative kinetics of urinary NGAL in neonates and to identify the threshold for accurate prediction of severe AKI requiring RRT in neonates and infants undergoing cardiac surgery with cardiopulmonary bypass.

The study is entirely observational, the decision to initiate RRT continues to be based on clinical evidence of fluid overload, low cardiac output and oliguria. Urine samples are collected during the early postoperative period, stored, than NGAL concentrations are measures on the ARCHITECT platform.

ELIGIBILITY:
Inclusion criteria :

* term neonates and infants undergoing heart surgery with cardiopulmonary bypass
* parents received written information

Exclusion criteria :

* preoperative documented kidney injury
* parents not informed, opposed

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: heterogeneous populations of children undergoing cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
NGAL kinetics | from 2 hours to 48 hours
  describe the kinetics of urinary NGAL in neonates after open heart surgery

SECONDARY OUTCOMES:
Ngal Threshold | from 2 hours to 48 hours
  identify the threshold for accurate prediction of severe AKI requiring renal replacement therapy
NGAL Algorithm | from 2 hours to 48 hours
  Development of an algorithm combining early clinical and laboratory criteria (including urinary NGAL) for prevention of renal failure and/or its worsening, and for early initiation of RRT in neonates and infants after cardiac surgery
NGAL Biomarkers | from 2 hours to 48 hours
  Setup of a sample repository, which will allow to study future biomarkers of AKI

CONTACTS AND LOCATIONS:
Overall Officials: Mirela Bojan, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Necker Hospital, Paris, France

REFERENCES:
- [Background] Bennett M, Dent CL, Ma Q, Dastrala S, Grenier F, Workman R, Syed H, Ali S, Barasch J, Devarajan P. Urine NGAL predicts severity of acute kidney injury after cardiac surgery: a prospective study. Clin J Am Soc Nephrol. 2008 May;3(3):665-73. doi: 10.2215/CJN.04010907. Epub 2008 Mar 12. PMID 18337554
- [Background] Mishra J, Dent C, Tarabishi R, Mitsnefes MM, Ma Q, Kelly C, Ruff SM, Zahedi K, Shao M, Bean J, Mori K, Barasch J, Devarajan P. Neutrophil gelatinase-associated lipocalin (NGAL) as a biomarker for acute renal injury after cardiac surgery. Lancet. 2005 Apr 2-8;365(9466):1231-8. doi: 10.1016/S0140-6736(05)74811-X. PMID 15811456
- [Background] Haase M, Bellomo R, Devarajan P, Schlattmann P, Haase-Fielitz A; NGAL Meta-analysis Investigator Group. Accuracy of neutrophil gelatinase-associated lipocalin (NGAL) in diagnosis and prognosis in acute kidney injury: a systematic review and meta-analysis. Am J Kidney Dis. 2009 Dec;54(6):1012-24. doi: 10.1053/j.ajkd.2009.07.020. Epub 2009 Oct 21. PMID 19850388
- [Derived] Bojan M, Basto Duarte MC, Lopez V, Tourneur L, Vicca S, Froissart M. Low perfusion pressure is associated with renal tubular injury in infants undergoing cardiac surgery with cardiopulmonary bypass: A secondary analysis of an observational study. Eur J Anaesthesiol. 2018 Aug;35(8):581-587. doi: 10.1097/EJA.0000000000000782. PMID 29432378
- [Derived] Bojan M, Basto Duarte MC, Ermak N, Lopez-Lopez V, Mogenet A, Froissart M. Structural equation modelling exploration of the key pathophysiological processes involved in cardiac surgery-related acute kidney injury in infants. Crit Care. 2016 Jun 5;20(1):171. doi: 10.1186/s13054-016-1350-1. PMID 27262736
- [Derived] Bojan M, Vicca S, Lopez-Lopez V, Mogenet A, Pouard P, Falissard B, Journois D. Predictive performance of urine neutrophil gelatinase-associated lipocalin for dialysis requirement and death following cardiac surgery in neonates and infants. Clin J Am Soc Nephrol. 2014 Feb;9(2):285-94. doi: 10.2215/CJN.04730513. Epub 2013 Nov 21. PMID 24262504